CLINICAL TRIAL: NCT07363642
Title: TAPER: A Prospective, Interventional, Multicentre, Single-Arm, Phase 3b Study to Evaluate the Step-Down of Maintenance Therapy in Patients With Severe Asthma Treated With Tezepelumab
Brief Title: Phase 3b Study in Patients With Severe Asthma Treated With Tezepelumab
Acronym: TAPER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5180L00021
Record Dates: First submitted 2025-11-25; First posted 2026-01-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Severe Asthma
Keywords: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tezepelumab (Experimental): Severe asthma taking medium-high dose ICS/LABA with up to one additional controller will be enrolled into this single arm treatment
  Interventions: Drug: Tezepelumab

INTERVENTIONS:
Drug: Tezepelumab — Severe asthma taking medium-high dose ICS/LABA with up to one additional controller will be enrolled into this single arm treatment

SUMMARY:
This study aims to explore the potential for Tezepelumab-treated severe asthmatic patients to effectively and safely reduce their background maintenance medication while maintaining asthma symptom control.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm Phase 3b study designed to evaluate the potential and safety of stepping down background maintenance therapy following the initiation of Tezepelumab treatment in Chinese patients with maintenance of asthma control.

This study will be conducted at approximately 70 study sites in China. The study duration for each patient will be up to 52 weeks. Approximately 400 patients with severe asthma taking medium-high dose ICS/LABA with/without LTRAs, LAMAs or theophylline will be enrolled into this single arm study.

ELIGIBILITY:
Inclusion Criteria:

1．Provision of informed consent prior to any study-specific procedures. Written informed consent, and assent when applicable for study participation must be obtained prior to any study related procedures being performed (local regulations are to be followed in determining the assent/consent requirements for children and parent[s]/guardian[s]) and according to international guidelines and/or applicable local guidelines.

Age 2. Patient must be aged 12-80 years old, inclusively, at the time of Visit 1(Week -1 to Week 0) For those patients, who are 17 on the day of Visit 1(Week -1 to Week 0) but will turn 18 after this day, will be considered an adolescent for the purposes of this study.

Type of Patient and Disease Characteristics 3. Documented history of physician-diagnosed asthma prior to Visit 1

* Documented post-bronchodilator (post-BD) reversibility in FEV1 of ≥12% and ≥200 mL in FEV1, or FEV1≥400 mL variability over time, or positive result of branchial provocation test within 12 months prior to Visit 1. If historical documentation is not available, reversibility must be demonstrated and documented at Visit 1.

  4. Documented current maintenance treatment with MD/HD ICS + LABA with up to one additional controller
* Other acceptable asthma controller includes LTRA, LAMA or theophylline 5. On stable MD/HD ICS (>250μg fluticasone propionate dry powder formulation equivalents total daily dose) + LABA stable for ≥2 months prior to enrollment 6. On stable LTRA or LAMA or theophylline (≥2 weeks) is allowed 7. Documented ACQ-5 ≥ 1.5 in Visit 1 8. Documented at least one exacerbation in the year prior to enrolment
* A qualifying historical asthma exacerbation is a symptomatic worsening requiring systemic corticosteroid (i.e., oral, intravenous (IV) or intramuscular; any healthcare setting or temporary increase from a stable maintenance dose of oral corticosteroid) or that resulted in hospitalization or emergency room/urgent care visit.
* Source documentation is required for physician-diagnosed asthma, ICS-LABA use and asthma exacerbations over the prior year. A patient verbal history suggestive of asthma symptoms and/or prior asthma exacerbations, but without supporting documentation, is not sufficient to satisfy these inclusion criteria.
* Examples of acceptable documentation of the asthma disease state and prior asthma exacerbations include clinic visit (primary or specialist Health care provider (HCP)), emergency room/urgent care, or hospital records listing asthma as a current problem, plus documentation of at least 1 asthma exacerbations during the 12 months prior to ICF.

Weight 9. Weight of ≥40 kg at Visit 1. Sex and Contraceptive/Barrier Requirements 10. Male and/or female Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Female patients:

* Females not of childbearing potential are defined as females who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Females will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to Visit 1(Week -1 to Week 0) without an alternative medical cause. The following age-specific requirements apply:
* Females < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and FSH levels in the postmenopausal range.
* Females ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.
* Female patients of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Females of childbearing potential who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control, as defined below, from enrolment throughout the study and until at least 8 weeks after last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician.
* The following are not acceptable methods of contraception: periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea. Female condom and male condom should not be used together.
* All WOCBP must have a negative serum pregnancy test result at Visit 1(Week -1 to Week 0).
* Highly effective birth control methods include: Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the patient (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments) [(periodic abstinence eg, calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to study intervention, and withdrawal are not acceptable methods of contraception], a vasectomised partner, Implanon®, bilateral tubal occlusion, intrauterine device/levonorgestrel intrauterine system, Depo-Provera™ injections, oral contraceptive, and Evra Patch™, Xulane™, or NuvaRing®.

Exclusion Criteria:

Medical Conditions

1. Unable to commit to the scheduled visits as required by the protocol, or unable to commit to undergoing protocol guided reductions in asthma therapy, as directed by the Investigator.
2. Clinically important pulmonary disease other than asthma (e.g., active lung infection, chronic obstructive pulmonary disease [COPD], bronchiectasis, pulmonary fibrosis, cystic fibrosis), or ever been diagnosed with pulmonary or systemic disease, other than asthma, that is associated with elevated peripheral eosinophil counts (e.g., allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).

   • Within the 12 months prior to Visit 1, a CT scan is required to exclude related diseases.
3. Current smokers at Visit 1 are not allowed. Former smokers with smoking history ≥ 10 pack-years at Visit 1 are not allowed; Former smokers with a smoking history of <10 pack years must have stopped for at least 6 months to be eligible.
4. History of alcohol or drug abuse within 12 months prior to Visit 1(Week -1 to Week 0).
5. A helminth parasitic infection diagnosed within 24 weeks prior to Visit 1(Week -1 to Week 0) that has not been treated with, or has failed to respond to, standard of care therapy.
6. History of anaphylaxis to any biologic therapy.
7. Known history of allergy or reaction to any component of the study treatment formulation.
8. Respiratory exacerbation requiring use of Systemic corticosteroids (SCS) or acute upper/lower respiratory infection that required antibiotics or antiviral medication within 30 days prior to Visit 1(Week -1 to Week 0). An extension of the screening period up to 3 months is allowed to ensure that a patient recovering from any repiratory exacerbation or acute upper/lower respiratory infection can be included.
9. A history of known immunodeficiency disorder, including human immunodeficiency virus.
10. Current or history of malignancy within 5 years before the screening visit with the following exceptions:

    * In-situ carcinoma of the cervix where curative therapy has been completed and patients are in remission for at least 12 months prior to screening.
    * Basal cell or superficial squamous skin cancer.
    * Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.
11. Exclusion for any of the following:

    * Previous allogeneic bone marrow transplant.
    * Non-leucocyte depleted whole blood transfusion within 120 days of genetic sample collection.
12. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

    1. Affect the safety of the patient throughout the study,
    2. Confound the study results or impact the scientific validity of the data outcome,
    3. Impede the patient's ability to complete the entire duration of study. Prior/Concomitant Therapy
13. Oral corticosteroid use during 4 weeks prior to Visit 1(Week -1 to Week 0).
14. Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, or any experimental anti-inflammatory therapy) within 3 months or 5 halflives (whichever is longer) prior to the date informed consent is obtained.
15. Receipt of any marketed or investigational biologic agent within 4 months or 5 half lives (whichever is longer) prior to Visit 1(Week -1 to Week 0) or receipt of any investigational non biologic agent within 30 days or 5 half-lives (whichever is longest) prior to Visit 1(Week -1 to Week 0). Exception:

    1. For marketed non-respiratory biologics, it is allowed if the patient is stable on treatment for at least 3 months prior to Visit 1(Week -1 to Week 0) and throughout the study.
    2. Covid-related prevention and treatment
16. Receipt of live attenuated vaccines 30 days prior to the date of first dose of Tezepelumab.
17. Intention to use any concomitant medication that is not permitted or failure to complete the required washout period for a particular prohibited medication.
18. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
19. Received bronchial thermoplasty (BT) as treatment of asthma within 12 months prior to Visit 1.
20. Received treatment with traditional Chinese herbs or proprietary Chinese medicines that have anti-asthmatic effects (excluding topical Chinese herbs) within 4 weeks prior to Visit 1 (Week -1 to Week 0) Prior/Concurrent Clinical Study Experience
21. Concurrent participation in another clinical study with an Investigational Product or a post-authorization safety study

    Diagnostic Assessments
22. Any clinically significant abnormal findings in physical examination, medical history, vital signs, haematology, or clinical chemistry during the enrolment period, which in the opinion of the investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete the entire duration of the study, e.g. HBV, HCV, active liver disease, Receipt of live attenuated vaccines 30 days prior to the date of visit 1.

    Other Exclusions
23. For females only - currently pregnant (confirmed with positive pregnancy test), breast-feeding, or lactating.
24. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
25. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
26. Previous enrolment in the present study.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2027-08-07 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the potential for Tezepelumab treated patients to reduce their standard of care asthma controller regimen in the overall patient population while maintaining asthma control | within 36 weeks after the first administration
  Main Endpoints: Proportion of patients with at least one controller medication category reduction at the end of reduction phase (week 36) while sustaining asthma control
  * discontinuation of LTRA, or
  * discontinuation of LAMA, or
  * discontinuation of theophylline, or
  * Reduce inhale therapy to MD ICS/LABA, or
  * Reduce inhale therapy to LD ICS/LABA
To assess the potential for Tezepelumab treated patients to reduce their standard of care asthma controller regimen in the overall patient population while maintaining asthma control | within 36 weeks after the first administration
  Supportive outcomes:
  * Proportion of patients with individual category reduction at end of reduction phase
  * Proportion of patients with ≥2 category reductions in controller medication

SECONDARY OUTCOMES:
To assess standard asthma efficacy measures for Tezepelumab treated patients for pulmonary function measured by pre-BD FEV1 | From week0~week48
  Change in pre-BD FEV1 measured in litres from:
  * Week 0 to week 1
  * week 0 to week 12 (beginning of induction phase to begining of reduction phase )
  * week 12 to week 36 (beginning of reduction phase to beginning of maintenance phase)
  * week 36 to week 48 (beginning of maintenance phase to the end of maintenance phase)
To assess standard asthma efficacy measures for Tezepelumab treated patients for asthma symptoms control measured by Asthma Control Questionnaire-5(ACQ-5) score | From week0~week48
  Change in measured by Asthma Control Questionnaire-5(ACQ-5) score from:
  * Week 0 to week 1
  * week 0 to week 12 (beginning of induction phase to begining of reduction phase )
  * week 12 to week 36 (beginning of reduction phase to beginning of maintenance phase)
  * week 36 to week 48 (beginning of maintenance phase to the end of maintenance phase) [ACQ-5: score 0-6, 6 means worse outcome]
To assess standard asthma efficacy measures for Tezepelumab treated patients for asthma symptoms control measured by St. George's Respiratory Questionnaire (SGRQ) score | From week0~week48
  Change in measured by St. George's Respiratory Questionnaire (SGRQ) score from:
  * Week 0 to week 1
  * week 0 to week 12 (beginning of induction phase to begining of reduction phase )
  * week 12 to week 36 (beginning of reduction phase to beginning of maintenance phase)
  * week 36 to week 48 (beginning of maintenance phase to the end of maintenance phase) [SGRQ: score 0-100, 100 means worse outcome]
To assess standard asthma efficacy measures for Tezepelumab treated patients for asthma symptoms control measured by Cough Evaluation Test (CET) score | From week0~week48
  Change in measured by Cough Evaluation Test (CET) score from:
  * Week 0 to week 1
  * week 0 to week 12 (beginning of induction phase to begining of reduction phase )
  * week 12 to week 36 (beginning of reduction phase to beginning of maintenance phase)
  * week 36 to week 48 (beginning of maintenance phase to the end of maintenance phase) [CET: score 5-25, 25 means worse outcome]
To assess if reductions in background therapies achieved at the end of reduction phase are maintained until the end of maintenance phase | From week36~week48
  Proportion of patients at the end of the maintenance phase(week48) who use the same background therapy that they achieved at the end of the reduction phase(week36)
To assess the proportion of patients achieving improvement in patient reported outcomes measured by ACQ-5 score for Tezepelumab treated patients | From week0~week52
  · Proportion of patients achieving ACQ-5 MCID score improvement (defined as change in ACQ-5 score≥-0.5 compared to week0 beginning of induction phase) [ACQ-5: score 0-6, 6 means worse outcome]
To assess overall asthma exacerbation rate during the study of severe asthma patients treated with Tezepelumab | from week0~week52
  • Annualized asthma exacerbation rate during the study (from first dose to EOT)
  Annualized asthma exacerbation rate Defined as Number of exacerbations×365.25/(Follow-Up Date-First Benralizumab dose date+1)
To assess biomarkers of severe asthma patients treated with Tezepelumab in the overall patient population | From week0~week52
  Baseline and follow-up visits, and change from baseline:
  • Blood EOS measured as cells per litre
To assess biomarkers of severe asthma patients treated with Tezepelumab in the overall patient population | From week0~week52
  Baseline and follow-up visits, and change from baseline:
  • FeNO measured as parts per billion
To assess biomarkers of severe asthma patients treated with Tezepelumab in the overall patient population | From week0~week52
  Baseline and follow-up visits, and change from baseline:
  • Total IgE measured as IU units per ml
To assess the potential for Tezepelumab Treated participants to obtain fast symptom control measured by Daily Diary questionnaire | from week0~week2
  • Change in daily rescue medication use times from baseline to week 2
To assess the change from baseline in nasal symptoms in severe asthma patients with comorbid CRSwNP measured by Sinonasal outcome test-22 (SNOT-22) score treated with Tezepelumab | from week0~week48
  Change in Sinonasal outcome test-22 (SNOT-22) score from beginning of week0(induction phase) to end of week48(maintenance phase) [SNOT-22: score 0-110, 110 means worse outcome]
To assess the potential for Tezepelumab Treated participants to obtain fast symptom control measured by Daily Diary questionnaire | from week0~week2
  • Percentage of nights with awakenings requiring rescue medication use times at week 2
To assess the potential for Tezepelumab Treated participants to obtain fast symptom control measured by lung function measured by PEF measured by liters per minute improvement | from week0~week2
  • Change in morning PEF measured as liters per minute from baseline to week 2
To assess the potential for Tezepelumab Treated participants to obtain fast symptom control measured by lung function measured by PEF measured by liters per minute improvement | from week0~week2
  • Proportion of patients reach clinically meaningful improvement in morning PEF measured as liters per minute (defined as 25 L/min) at week 2
To assess the proportion of patients achieving improvement in lung function measured by pulmonary function measured by pre-BD FEV1 measured in litres for Tezepelumab treated patients | From week0~week52
  • Proportion of patients achieving pre-FEV1 MCID measured in litres improvement (defined as patients who achieve either a ≥ 5% or ≥ 100 mL improvement compared to week0 beginning of induction phase)
To assess the proportion of patients achieving improvement in patient reported outcomes measured by SGRQ score for Tezepelumab treated patients | From week0~week52
  · Proportion of patients achieving SGRQ MCID score improvement (defined as change in SGRQ score≥-4 compared to week0 beginning of induction phase) [SGRQ: score 0-100, 100 means worse outcome]
To assess the proportion of patients achieving improvement in patient reported outcomes measured by CET score for Tezepelumab treated patients | From week0~week52
  • Proportion of patients achieving CET MCID score improvement (defined as change in CET score≥2 compared to week0 beginning of induction phase) [CET: score 5-25, 25 means worse outcome]

CONTACTS AND LOCATIONS:
Overall Officials: KeFang Lai, Professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; FengMing Luo, Professor, Principal Investigator — Sichuan University West China Hospital
Locations (44):
- China (44):
  - Research Site, Beijing
  - Research Site, Binzhou
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Deyang
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jiangmen
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Leshan
  - Research Site, Linyi
  - Research Site, Luzhou
  - Research Site, Meizhou
  - Research Site, Mianyang
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Quanzhou
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining Shi
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Zhangzhou
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
  - Research Site, Zhongshan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, it indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/